CLINICAL TRIAL: NCT04514302
Title: Phase I, Randomized, Placebo-controlled, Double-blind, Study to Evaluate the Safety and Antiviral Efficacy of Three Different Single Doses of Anti-SARS-CoV-2 Equine Antibody F(ab')2 Fragments (INOSARS) in Adult Patients With Mild COVID-19
Brief Title: Safety and Efficacy of Anti-SARS-CoV-2 Equine Antibody F(ab')2 Fragments (INOSARS) for Adult Patients With Mild COVID-19
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TecSalud Investigación Clínica (Other)
Collaborators: Inosan Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TS202101
Record Dates: First submitted 2020-08-12; First posted 2020-08-14 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: COVID-19
Keywords: COVID-19; SARS-CoV-2; Immunoglobulin fragments; Hyperimmune equine serum; Passive immunotherapy
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Parallel
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Single dose of a 150 mL saline solution administered intravenously as an infusion over 40 min.
  Interventions: Drug: Placebo
- INOSARS dose 1 (Experimental): Single dose of 5 mg/kg in a 150 mL saline solution administered intravenously as an infusion over 40 min.
  Interventions: Drug: Anti-SARS-CoV-2 equine immunoglobulin F(ab')2 fragments (INOSARS)
- INOSARS dose 2 (Experimental): Single dose of 15 mg/kg in a 150 mL saline solution administered intravenously as an infusion over 40 min.
  Interventions: Drug: Anti-SARS-CoV-2 equine immunoglobulin F(ab')2 fragments (INOSARS)
- INOSARS dose 3 (Experimental): Single dose of 30 mg/kg in a 150 mL saline solution administered intravenously as an infusion over 40 min.
  Interventions: Drug: Anti-SARS-CoV-2 equine immunoglobulin F(ab')2 fragments (INOSARS)

INTERVENTIONS:
Drug: Placebo — Placebo of saline solution of equal volume and infusion. Content of the infusion bag and tubing will be concealed with opaque covering.
  Other Names: Control
  Arms: Placebo
Drug: Anti-SARS-CoV-2 equine immunoglobulin F(ab')2 fragments (INOSARS) — INOSARS is a polyvalent passive immunization based on anti-SARS-CoV-2 immunoglobulin F(ab')2 fragments from hyperimmune equine serum. Inactive ingredients: water for injection, sodium chloride and less than 10% of total protein content.
  Other Names: INOSARS
  Arms: INOSARS dose 1; INOSARS dose 2; INOSARS dose 3

SUMMARY:
This is a randomized, placebo-controlled, double-blind phase I clinical study of anti-SARS-CoV-2 equine immunoglobulin F(ab')2 fragments (INOSARS) to evaluate the safety and antiviral efficacy for the treatment of adult patients with mild COVID-19 and low risk of disease progression.

ELIGIBILITY:
Key Inclusion criteria

* Outpatient with a RT-qPCR confirmation of SARS-CoV-2 infection
* Body Mass Index (BMI) at screening of 18.0 - 34.9 kg/m^2
* Presence of at least one symptom consistent with COVID-19
* Mild illness as defined by no requirement of supplementary oxygen or hospitalization criteria are met

Key Exclusion criteria

* Presence of a risk factor for disease progression documented for COVID-19 such as: uncontrolled diabetes, uncontrolled hypertension, cardiovascular disease, pulmonary disease, COPD, asthma, active cancer, immunosuppression, hypercoagulable states, CKD currently under dialysis
* Documented allergy to equine serum proteins
* Previous hospitalization due to COVID-19
* Supplementary oxygen, invasive ventilation, or mechanical circulatory support requirements
* Having received convalescent plasma or intravenous immunoglobulins for the treatment of COVID-19
* Previous vaccination or plans to get vaccinated for COVID-19
* In the opinion of investigator, other health conditions that suppose an increased risk of progression of disease

NOTE: Other inclusion/exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2021-12-07 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Average change from baseline in viral load as quantified by RT-qPCR from nasopharyngeal swab samples | Baseline to days 2, 4, 7, 14 and 28
Proportion of patients with undetectable viral load as quantified by RT-qPCR from nasopharyngeal swab samples | At days 2, 4, 7, 14 and 28
Time of viral activity | Baseline to 28 days
  Number of days in which viral load remains detectable as quantified by RT-qPCR from nasopharyngeal swab samples

SECONDARY OUTCOMES:
Adverse events presented early after infusion | Baseline to 24 hrs
  Number of adverse events per group presented in the first 24 hours
Adverse events presented later after infusion | Day 2 until day 28
  Number of adverse events per group presented 24 hours past infusion
Incidence of anti-INOSARS antibodies | Baseline and day 28

CONTACTS AND LOCATIONS:
Overall Officials: José F Castilleja-Leal, MD, Principal Investigator — TecSalud Investigación Clínica
Locations (1):
- Hospital San José, Tec de Monterrey, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beigel JH, Tomashek KM, Dodd LE, Mehta AK, Zingman BS, Kalil AC, Hohmann E, Chu HY, Luetkemeyer A, Kline S, Lopez de Castilla D, Finberg RW, Dierberg K, Tapson V, Hsieh L, Patterson TF, Paredes R, Sweeney DA, Short WR, Touloumi G, Lye DC, Ohmagari N, Oh MD, Ruiz-Palacios GM, Benfield T, Fatkenheuer G, Kortepeter MG, Atmar RL, Creech CB, Lundgren J, Babiker AG, Pett S, Neaton JD, Burgess TH, Bonnett T, Green M, Makowski M, Osinusi A, Nayak S, Lane HC; ACTT-1 Study Group Members. Remdesivir for the Treatment of Covid-19 - Final Report. N Engl J Med. 2020 Nov 5;383(19):1813-1826. doi: 10.1056/NEJMoa2007764. Epub 2020 Oct 8. PMID 32445440